CLINICAL TRIAL: NCT00564863
Title: Strain and Dose-Finding Study of DS26-1 and WS0115A Enterotoxigenic E. Coli (ETEC) Challenge Strains That Express CS19 Fimbriae
Brief Title: Dose-Finding Study of CS19 Expressing ETEC Challenge Strains
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, August Louis Bourgeois, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIR 240; WIRB Approval Number 20071069 (Other: WIRB); Gm 100018 (Other Grant/Funding Number: Army)
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Travelers' Diarrhea
Keywords: Diarrhea; ETEC
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: This is a phase 1, open-label, strain and dose-finding study designed to establish a human challenge model for CS19-ETEC that causes a > 80% attack rate without causing high output diarrhea. This will be a strain and dose-finding study in which CS19-ETEC strain WS0115A will be administered at a starting inoculum of 5 x 108 colony forming units (cfu) to 5 subjects as the initial step to establish a human disease model. If an 80% attack rate (AR) for predefined diarrheal disease is achieved without high output diarrhea, the same inoculum will be given to 5 - 10 more subjects for confirmation of AR. If an 80% AR is not achieved, AR and severity of disease will be evaluated to determine if the dose should be increased. The same sequence may be conducted with DS26-1 as necessary.
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS19 expressing ETEC strain (Other): Ascending dose finding study in 5-10 subjects per dose; to identify the dose able to give a diarrheal attack rate greater than or equal to 80%.
  Interventions: Biological: CS19 expressing ETEC strain

INTERVENTIONS:
Biological: CS19 expressing ETEC strain — Wild type ETEC strain expressing the colonization faction CS19, and LT and ST enterotoxins.

SUMMARY:
This will be a strain and dose-finding study in which CS19-ETEC strain WS0115A will be administered at a starting inoculum of 5 x 108 colony forming units (cfu) to 5 subjects as the initial step to establish a human disease model. If an 80% attack rate (AR) for predefined diarrheal disease is achieved without high output diarrhea, the same inoculum will be given to 5 - 10 more subjects for confirmation of AR. If an 80% AR is not achieved, AR and severity of disease will be evaluated to determine if the dose should be increased. The same sequence may be conducted with DS26-1 as necessary. If the WS0115A strain causes high output diarrhea, the dose will be adjusted down and further dose characterization continued. An iterative process will be used to select the optimal strain and dose with each step reviewed and approved by the medical monitor.

DETAILED DESCRIPTION:
This is a phase 1, open-label, strain and dose-finding study designed to establish a human challenge modelfor CS19-ETEC that causes a > 80% attack rate without causing high output diarrhea. This study design is identical to that of the CS17 challenge model recently completed. Two strains of CS19-ETEC isolated from human diarrheal cases have been identified and characterized. Each clinical isolate was used to generate a cGMP MCB and procedures were established to create a fresh inoculum to administer orally in a sodium bicarbonate solution for challenge. Refer to Section 8 for full details on the isolation and preparation of these strains.

CS19-ETEC strain WS0115A (toxin phenotype of LT+ ST+ and serotype O114:H-) will be the lead strain and will be administered orally to an initial cohort of 5 subjects. This strain was isolated from the stool of a 12-month-old Egyptian girl suffering from watery diarrhea identified during a surveillance study conducted in Abees, Egypt from 1993 to 1995 by investigators at the Naval Medical Research Unit-3 (NAMRU-3), Cairo, Egypt. A negative microbiologic work-up for copathogens (other bacterialenteropathogens, rotavirus, Giardia lamblia, Entamoeba histolytica, and Cryptosporidium) supports that the isolated WS0115A strain was pathogenic in this child. Since this strain has an LT+ST+ toxin phenotype, it is the preferred strain to lead in testing the challenge model, since heterologous protection by bovine milk IgG anti-CsbD against an LT+ST+ phenotype would offer a more robust test of the protection afforded by anti-colonization. The alternate strain, CS-19 ETEC strain DS26-1 (toxin phenotype LT+ST-;serotype O8:H9) was isolated in 1990 at the U.S. Navy Forward Laboratory from a U.S. soldier with diarrhea while on deployment to Saudi Arabia during Operation Desert Shield. A negative microbiologic work-up for copathogens (Salmonella typhi, Vibrio cholerae, Giardia lamblia or Entamoeba histolytica)supports that the isolated DS26-1 strain was pathogenic in this individual. Each clinical isolate was used to generate a cGMP master cell bank and procedures were established to create a fresh inoculum to administer orally in a sodium bicarbonate solution for challenge. Refer to Section 8 for full details on the isolation and preparation of these strains.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 45 years of age, inclusive.
2. General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by principal investigator (PI) or PI in consultation with the medical monitor and Sponsor.
3. Demonstrate comprehension of the protocol procedures and knowledge of ETEC illness by passing a written examination (pass grade ≥ 70%)
4. Willing to participate after informed consent obtained.
5. Available for entire inpatient portion of study and all outpatient study visits.
6. Negative serum pregnancy test at screening (initial visit and day -7 to - 3) and a negative urine pregnancy test on the day of admission to the inpatient phase for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Alternatively, abstinence alone is acceptable. Female subjects who are unable to bear children must provide supporting documentation (e.g., prior tubal ligation or hysterectomy).

Exclusion Criteria:

1. Presence of a significant medical condition, (e.g., psychiatric conditions or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease, alcohol or illicit drug abuse/dependency), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
2. Immunosuppressive illness or IgA deficiency (below the normal limits)
3. Positive serology results for HIV, HBsAg, or HCV antibodies.
4. Significant abnormalities in screening laboratory hematology, serum chemistry, urinalysis, as determined by PI or PI in consultation with the medical monitor and Sponsor.
5. Allergy to fluoroquinolones, cotrimoxazole, or ampicillin/penicillin (excluded if allergic to two of three).
6. Fewer than 3 stools per week or more than 3 stools per day as the usual frequency; loose or liquid stools other than on an occasional basis.
7. History of diarrhea in the 2 weeks prior to planned inpatient phase.
8. Regular use of laxatives or any agent that increases gastric pH (regular defined as at least weekly).
9. Use of antibiotics during the 7 days before bacterial dosing or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing.
10. Travel to countries where ETEC or cholera infection is endemic (most of the developing world) within two years prior to dosing.
11. History of vaccination for or ingestion of ETEC, cholera, or LT toxin.
12. Stool culture (collected no more than 1 week prior to admission) positive for ETEC or other bacterial enteric pathogens (Salmonella, Shigella and Campylobacter).
13. Use of any investigational product within 30 days preceding the receipt of the challenge inoculum, or planned use during the active study period.
14. Use of any medication known to affect the immune function (e.g., corticosteroids) within 30 days preceding receipt of the challenge inoculum or planned use during the active study period. (Topical and intra-articular steroids will not exclude subjects). MANAGEMENT

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-09-04 (Actual)

PRIMARY OUTCOMES:
Develop of diarrhea. | 120 hours after challenge

SECONDARY OUTCOMES:
Development of moderate to severe diarrhea | 120 hours after challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robin McKenzie, M.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research - Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - General Clinical Research Center of the Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No